CLINICAL TRIAL: NCT07119346
Title: Effect of Ultrasound-guided External Oblique Intercostal Fascial Plane Block in Pediatric Patients Undergoing Laparoscopic Gastrostomy: A Prospective Randomized Controlled Trial
Brief Title: EOI Block for Laparoscopic Gastrostomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2505-109-1643
Record Dates: First submitted 2025-08-11; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Gastrostomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOI block group (Experimental)
  Interventions: Procedure: EOI block
- control group (Sham Comparator)
  Interventions: Procedure: sham block

INTERVENTIONS:
Procedure: EOI block — EOI block with 0.25% ropivacaine 1 mL/kg (max 40 mL) bilaterally under ultrasound guidance
  Arms: EOI block group
Procedure: sham block — Sham block with equal volume of normal saline bilaterally under ultrasound guidance
  Arms: control group

SUMMARY:
This randomized controlled trial will evaluate the efficacy of ultrasound-guided external oblique intercostal fascial plane (EOI) block in reducing intraoperative and postoperative pain in pediatric patients undergoing laparoscopic gastrostomy under general anesthesia. Forty patients aged 3-18 years will be randomly allocated to receive either bilateral EOI block with 0.25% ropivacaine or sham block with normal saline. Primary outcome is percent change in heart rate at surgical incision. Secondary outcomes include intraoperative fentanyl use, perioperative analgesic requirements, postoperative pain scores (r-Face, Legs, Activity, Cry, Consolability(r-FLACC) and Pediatric Pain Profile), Analgesia Nociception Index values, and analgesia-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for laparoscopic gastrostomy at Seoul National University Children's Hospital

Age ≥3 and <18 years

Exclusion Criteria:

* Unstable vital signs

Contraindications to ropivacaine or opioids

Severe hepatic or renal dysfunction

Other investigator-determined ineligibility

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Percent change in heart rate at surgical incision | At surgical incision (baseline immediately before incision and within 10 minutes after incision).
  Post-incision HR - Pre-incision HR) / Pre-incision HR × 100

SECONDARY OUTCOMES:
Intraoperative fentanyl use | From induction of anesthesia to end of surgery.
Percent change in mean arterial pressure at incision | At surgical incision (baseline immediately before incision and within 10 minutes after incision).
Intraoperative max-min heart rate | Intraoperative period (skin incision to end of surgery).
Intraoperative max-min mean arterial pressure | Intraoperative period (skin incision to end of surgery).
ANI time-weighted average outside target (50-80) | From induction of anesthesia to end of anesthesia (arrival to PACU).
r-Face, Legs, Activity, Cry, Consolability pain scores | At PACU 15 minutes and 30 minutes; and at 1, 3, 6, and 24 hours after surgery.
Pediatric Pain Profile score | 24 hours after surgery.
analgesia nociception index (ANIm) values in PACU | At 15 and 30 minutes after PACU arrival.
Non-opioid analgesic consumption (mg/kg) | From end of surgery to 24 hours postoperatively.
Opioid analgesic consumption (mcg/kg) | From end of surgery to 24 hours postoperatively.
Analgesic-related adverse effects | Up to 24 hours after surgery.
  nausea, vomiting, pruritus

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea